CLINICAL TRIAL: NCT02355054
Title: Detecting Recurrent Prostate Cancer With C-11 Choline Positron Emission Tomography: An Expanded Access Study
Status: Approved for marketing | Type: Expanded Access
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Farrokh Dehdashti, Professor of Radiology, Washington University School of Medicine
Other Study IDs: 201411142
Record Dates: First submitted 2015-01-29; First posted 2015-02-04 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Cancer of the Prostate
Keywords: Recurrent
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

INTERVENTIONS:
Drug: C-11 Choline PET Imaging — Patients will receive IV injection of C-11 Choline followed by imaging from the base of the brain to the upper thigh on a PET/CT or a PET/MRI scanner

SUMMARY:
The purpose of this study is to provide clinical access to PET/CT and PET/MRI with C-11 choline for evaluation of men with biochemically recurrent prostate cancer while awaiting approval of the Washington University Abbreviated New Drug Application for C-11 choline.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have biopsy-proven adenocarcinoma of the prostate initially treated with curative intent (surgery and radiation therapy are most common treatments but other treatments are also eligible).
2. Biochemical recurrence defined as any of the following:

   * PSA ≥ 0.2 ng/mL in at least two sequential tests for patients treated with surgery.
   * PSA ≥ 2.0 ng/mL above the post therapy nadir for patients treated with radiation therapy, brachytherapy or cryotherapy.
   * PSA ≥ 2.0 ng/ml above the most recent therapy nadir for patients who have received additional treatment in the recurrent setting.
3. Patient must have undergone standard-of-care restaging that does not clearly identify site(s) of active disease. Standard staging examinations may include one or more of the following: CT or MRI, bone imaging (either Tc-99m bisphosphonate scintigraphy or F-18 sodium fluoride PET), OR In-111 capromab pendetide scintigraphy.
4. Age > 18 years.
5. Patient must be able to tolerate PET/MRI or PET/CT imaging
6. Patient must be able to understand and willing to sign a written informed consent document.
7. Patient must be able to understand and willing to sign an Advance Beneficiary Notice (ABN) (Medicare patient) or a Notice of Non-coverage (NNC) from (non-Medicare patient) that addresses the potential cost to the patient of C-11 choline PET/CT or PET/MRI.

Exclusion Criteria:

1. For patients planned to have PET/MRI:

   * Patient must not have claustrophobia or any other contraindication to MRI as evaluated by a standardized MRI safety questionnaire.
   * If applicable, patient must not have renal insufficiency (estimated glomerular filtration rate < 30 mL/min/1.73 m2 based on measurement within the past 60 days) or be undergoing dialysis as these conditions preclude safe administration of MRI contrast agents. NOTE: At the discretion of principal investigator, a subject may be allowed to enroll/continue on study and undergo imaging without the administration of contrast in the event of renal insufficiency.
   * If applicable, patient must not have a known prior reaction to gadolinium based MRI contrast agents.
2. For patients planned to have PET/CT:

   * Patient must not have claustrophobia that would preclude PET/CT imaging or other contraindications to CT imaging.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, Barnes-Jewish Hospital, St Louis, Missouri, United States